CLINICAL TRIAL: NCT01029847
Title: Adalimumab in Axial Spondyloarthritis. An Investigation of Whole-body MRI, MRI of Sacroiliac Joints and Spine and Soluble Biomarkers of Joint Inflammation and Damage.
Brief Title: Adalimumab in Axial Spondyloarthritis (ASIM) - MRI and Biomarkers in Patients With Spondyloarthritis
Acronym: ASIM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Professor Mikkel Østergaard, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASIM
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Spondyloarthritis
Keywords: Patients with axial spondyloarthritis
MeSH Terms: conditions — Spondylarthritis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Adalimumab (Active Comparator): TNF-alpha inhibitor
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Sc. inj. adalimumab 40 mg every other week for 42 to 48 weeks. At week 24, clinical non-responders (not fulfilling primary outcome measure) were allowed treatment with other drugs, following local treatment guidelines.
  Arms: Adalimumab
Drug: Placebo — sc. inj. placebo every other week, week 0, 2, and 4. Sc. inj. adalimumab 40 mg every other week from week 6.
  At week 24, clinical non-responders (not fulfilling primary outcome measure) were allowed treatment with other drugs, following local treatment guidelines.
  Arms: Placebo

SUMMARY:
Investigation of wholebody MRI and circulating biomarkers of inflammation, cartilage and bone metabolism in patients with spondyloarthritis treated with adalimumab. Furthermore to compare ultrasound examination with wholebody MRI etc.

ELIGIBILITY:
Inclusion Criteria:

* Spondyloarthritis (SpA) according to the new ASAS criteria for axial SpA
* BASDAI > 40 mm despite NSAIDs
* Clinical indication for treatment with TNF-alpha inhibitor
* Age > 18 years old and < 85 years old
* Sufficient contraception for women
* Capable of giving informed consent
* Capable of complying with the examination program of the protocol

Exclusion Criteria:

* Pregnancy wish, pregnancy or breast-feeding
* DMARDs within 4 weeks prior to inclusion
* Oral, intra-articular or intramuscular glucocorticoid within 4 weeks prior to inclusion
* The use of other study drugs within 4 weeks prior to inclusion or less than 5 half-lives of the study drug before inclusion if this is more than 4 weeks
* The use of suspected disease-modifying or immunosuppressive drugs within 4 weeks prior to inclusion
* DMARDs are allowed during the study, but the dose cannot be changed from 4 weeks prior to inclusion through week
* Contraindications for TNF-α inhibitor treatment
* Contraindications for MRI
* Known recent drug or alcohol abuse
* Failure to provide written consent
* Incapable of complying with the examination program for physical or mental reasons

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) of 20 mm or 50% | 24 weeks

SECONDARY OUTCOMES:
Number of peripheral and axial joints and entheses with inflammation, circulating biomarkers of inflammation, cartilage and bone metabolism, conventional clinical parameters and changes in these during treatment with adalimumab. | 24 week

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Østergaard, Professor, Principal Investigator — Dep. of Rheumatology, Glostrup Hospital; Susanne J Pedersen, MD, Study Chair — Dep. of Rheumatology, Glostrup Hospital; Inge J Sørensen, Study Chair — Dep. of Rheumatoogy, Glostrup Hospital
Locations (8):
- Denmark (8):
  - Dep. of medicine, Herlev Hospital, Copenhagen
  - Dep. of Radiology, Herlev Hospital, Copenhagen
  - Dep. of Rheumatology, Frederiksberg and Bispebjerg Hospitals, Copenhagen
  - Dep. of Rheumatology, Gentofte Hospital, Copenhagen
  - Dep. of Rheumatology, Hvidovre Hospital, Copenhagen
  - Dep. of Rheumatologym Glostrup Hospital, Copenhagen
  - Dep. of Rheumatology, Helsinør Hospital, Hørsholm
  - Dep. of Rheumatology, Køge Hospital, Køge

REFERENCES:
- [Derived] Krabbe S, Eshed I, Sorensen IJ, Jensen B, Moller JM, Balding L, Madsen OR, Pedersen SJ, Ostergaard M. Whole-body Magnetic Resonance Imaging Inflammation in Peripheral Joints and Entheses in Axial Spondyloarthritis: Distribution and Changes during Adalimumab Treatment. J Rheumatol. 2020 Jan;47(1):50-58. doi: 10.3899/jrheum.181159. Epub 2019 Apr 1. PMID 30936290
- [Derived] Krabbe S, Sorensen IJ, Jensen B, Moller JM, Balding L, Madsen OR, Lambert RGW, Maksymowych WP, Pedersen SJ, Ostergaard M. Inflammatory and structural changes in vertebral bodies and posterior elements of the spine in axial spondyloarthritis: construct validity, responsiveness and discriminatory ability of the anatomy-based CANDEN scoring system in a randomised placebo-controlled trial. RMD Open. 2018 Mar 16;4(1):e000624. doi: 10.1136/rmdopen-2017-000624. eCollection 2018. PMID 29556419